CLINICAL TRIAL: NCT00491153
Title: Sensitivity and Specificity of Aridol Challenge for a Diagnosis of Asthma by a Specialist Pulmonologist
Status: Terminated | Type: Observational
Why Stopped: due to low recruitment rate secondary to very stringent inclusion criteria
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 4.2006.3606(REK); 2006-006469-17 (Other: EUDRACT)
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: asthma; airway hyperresponsiveness; dry powder mannitol inhalation; methacholine
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to estimate the sensitivity, specificity and positive and negative predictive values of a positive Aridol challenge with respect to a specialist pulmonologist diagnosis of asthma in corticosteroid naive subjects with asthma-like symptoms and no previous diagnosis of asthma. The comparator is methacholine provocation

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Provisional or possible asthma diagnosis
* FEV1 at least 70% of predicted at inclusion

Exclusion Criteria:

* Contraindications for bronchial provocation challenge or spirometry
* Respiratory tract infection within previous 6 weeks
* Significant co-morbidity
* > 10 pack year smoking history
* Other lung diseases
* Pregnancy, lactation

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with a tentative diagnosis of asthma or suspected asthma referred to a pulmonologist for evaluation
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2007-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity and positive and negative predictive values of a positive Aridol bronchial challenge test | 1 day
  with respect to asthma diagnosis by a specialist pulmonary physician in corticosteroid-naïve subjects presenting with signs and symptoms suggestive of asthma but without a definitive diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ernst Omenaas, MD, PhD, Study Director — Haukeland University Hospital
Locations (3):
- Norway (3):
  - St.Olavs Hospital, University Hospital of Trondheim, Trondheim, South Trøndelag
  - Dr Alf Magne Heggli medical practice, Trondheim, South Trøndelag
  - Haukeland University Hospital, Bergen

REFERENCES:
- [Background] Anderson SD, Charlton B, Weiler JM, Nichols S, Spector SL, Pearlman DS; A305 Study Group. Comparison of mannitol and methacholine to predict exercise-induced bronchoconstriction and a clinical diagnosis of asthma. Respir Res. 2009 Jan 23;10(1):4. doi: 10.1186/1465-9921-10-4. PMID 19161635